CLINICAL TRIAL: NCT00071084
Title: An Open-Label Therapeutic Exploratory Clinical Trial of HuMax-CD4, a Fully Human Monoclonal Anti-CD4 Antibody, in Patients With Advanced Stage (IIA-IVB) Cutaneous T-cell Lymphoma
Brief Title: Clinical Trial of HuMax-CD4, a New Drug to Treat Advanced Stage T-Cell Lymphoma in the Skin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hx-CD4-008
Record Dates: First submitted 2003-10-10; First posted 2003-10-15 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: Skin cancer; Lymphoma; Mycosis fungoides; Sezary syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Skin Neoplasms; Lymphoma; Mycosis Fungoides; Sezary Syndrome | interventions — zanolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HuMax-CD4 280 milligrams (mg) (Experimental)
  Interventions: Drug: HuMax-CD4
- HuMax-CD4 980 mg (Experimental)
  Interventions: Drug: HuMax-CD4

INTERVENTIONS:
Drug: HuMax-CD4 — HuMax-CD4 280 mg was administered as a subcutaneous (SC) infusion once daily (OD) up to 16 weeks.
  Other Names: Zanolimumab
  Arms: HuMax-CD4 280 milligrams (mg)
Drug: HuMax-CD4 — HuMax-CD4 980 mg was administered as a SC infusion OD up to 16 weeks.
  Other Names: Zanolimumab
  Arms: HuMax-CD4 980 mg

SUMMARY:
The purpose of this trial is to determine the effect of HuMax-CD4, as a treatment for advanced stage (late stage) cutaneous T-cell lymphoma (CTCL). Almost all participants who are affected by late stage CTCL have many cancerous cells which bear a receptor called CD4. HuMax-CD4 is an investigational drug directed against this receptor. There is no placebo in this trial; all participants will be treated with HuMax-CD4. The response rates, duration of responses, relief of symptoms, and safety profile of HuMax-CD4 will be evaluated during this trial.

ELIGIBILITY:
Inclusion criteria

* Medical diagnosis of CTCL, and positivity for the CD4 receptor.
* Late stage CTCL.
* Have received at least one prior anti-cancer therapy with inadequate effect.
* World Health Organization (WHO) performance status 0,1 or 2

Exclusion Criteria

* Certain rare types of CTCL.
* Previous treatment with other anti-CD4 medications.
* More than two previous treatments with systemic chemotherapy.
* Certain anti-psoriasis or anti-cancer therapies within the last 4 weeks before entering this trial.
* Some types of steroid treatments less than two weeks before entering the trial.
* Prolonged exposure to sunlight or UV light during the trial.
* Other cancer diseases, except certain skin cancers or cervix cancer.
* Chronic infectious disease requiring medication.
* Certain serious medical conditions, including kidney or liver disease, some psychiatric illnesses, and stomach, lung, heart, hormonal, nerve or blood diseases.
* Pregnant or breast-feeding women.
* Women of childbearing age who are unable or unwilling to use an IUD or hormonal birth control during the whole trial.
* If you are participating in another trial with a different new drug 4 weeks before you enter this trial.

Note: Other protocol defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-05-27 (Actual); Primary Completion 2004-06-29 (Actual); Study Completion 2004-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved Complete and Partial Responses Assessed by Composite Assessment of Index Lesion Disease Severity (CA) Scale | Up to 20 weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Graded as per Severity | From Baseline (Day 0) up to end of study (Week 20)
Percentage of Participants With Physician's Global Assessment of Clinical Condition (PGA) Response | Up to 20 weeks
Percentage of Participants with Change from Baseline in Participant's Assessment of Pruritus Scale | Baseline, up to Week 20
  The participants were assessed pruritus on a 5-point scale from 0-4: 0. No complaint of itching on lesion; 1. Mild: Occasional transient itching on lesion; 2. Moderate: Frequent itching, every 1-3 hours; reflex scratching; 3. Severe: Compelling itching; interrupts daily activities; must be scratched; 4. Very severe: Unrelieved itching: prevents routine activities; awakens patient from sleep.
Time to Response | From first dose to achieving a response (up to approximately 12 weeks)
Response Duration | From achieving first response to last response/until relapse (up to approximately 22 weeks)
Time to Disease Progression | From first dose until disease progressed (Up to 16 weeks)
Percentage of Participants with Change From Baseline in Total Body Surface Area (BSA) | Baseline up to Week 21
Change from Baseline in Physician's Erythroderma Severity Assessment | Baseline, Week 20
Number of Participants With Positive Human Anti Human Antibodies (HAHA) Titres | Up to Week 20

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Stanford University Med Ctr., Dept of Dermatology, Stanford, California
  - University of Texas, M.D. Anderson Cancer Center, Houston, Texas
- Münster, Germany
- Stockholm, Sweden
- London, United Kingdom